CLINICAL TRIAL: NCT00294515
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study of the Efficacy and Safety of up to 100 Days of Valganciclovir Versus up to 200 Days of Valganciclovir for Prevention of Cytomegalovirus (CMV) Disease in High-Risk Kidney Allograft Recipients
Brief Title: IMPACT Study: A Study of Valcyte (Valganciclovir) for Prevention of Cytomegalovirus Disease (CMV) in Kidney Allograft Recipients
Acronym: IMPACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NT18435
Record Dates: First submitted 2006-02-21; First posted 2006-02-22 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Cytomegalovirus Infections
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valganciclovir up to 100 days (Experimental): Valganciclovir for up to 100 days post kidney transplant
  Interventions: Drug: Valganciclovir
- Valganciclovir up to 200 days (Active Comparator): Valganciclovir for up to 200 days post kidney transplant
  Interventions: Drug: Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — 900 mg orally daily for up to 100 days
  Other Names: Valcyte
  Arms: Valganciclovir up to 100 days
Drug: Valganciclovir — 900 mg orally daily for up to 200 days
  Other Names: Valcyte
  Arms: Valganciclovir up to 200 days

SUMMARY:
This study will determine the relative efficacy and safety of up to 100 days Valcyte prophylaxis relative to up to 200 days Valcyte prophylaxis when given for the prevention of CMV disease in high-risk (D+/R-) kidney allograft recipients. The anticipated time on study treatment is 3-12 months and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 16 years of age
* CMV seronegative recipient of primary or secondary renal allograft from a living or cadaveric seropositive donor
* Adequate hematological and renal function
* Patients and partners must agree to maintain effective birth control for 90 days following cessation of study medication

Exclusion Criteria:

* CMV disease, or receipt of anti-CMV therapy within 30 days prior to screening
* Multi-organ transplant recipient
* Hepatitis B, hepatitis C or HIV positive
* Women who are pregnant or lactating

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2006-03-31 (Actual); Primary Completion 2008-08-31 (Actual); Study Completion 2009-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (80):
- United States (23):
  - Uni of Alabama At Birmingham, Birmingham, Alabama
  - National Institute of Transplantation, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Ucsd Medical Center; Kidney Transplantation, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - Uni of California San Francisco; Transplant Services, San Francisco, California
  - Lifelink Healthcare Inst., Tampa, Florida
  - Rush-Presbyterian St. Luke'S Medical Center; Rush Uni Renal Transplant Program, Chicago, Illinois
  - Indiana Uni Medical Center; Surgery & Microbiology/Immunology, Indianapolis, Indiana
  - New England Medical Center; Division of Transplant Surgery, Boston, Massachusetts
  - Uni of Michigan Medical Center, Ann Arbor, Michigan
  - Uni of Minnesota Medical Center; Dept of Surgery, Minneapolis, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Barnabas Medical Center, Livingston, New Jersey
  - Robert Wood Johnson Uni Hospital; Anesthesia, New Brunswick, New Jersey
  - Wake Forest Uni School of Medicine; Section on Infectious Diseases, Winston-Salem, North Carolina
  - Oregon Health Sciences Uni ; Division of Nephrology, Portland, Oregon
  - Hahnemann Uni Hospital; Division of Transplant/Dept. of Surgery, Philadelphia, Pennsylvania
  - Uni of Pennslyvania Medical Center, Philadelphia, Pennsylvania
  - Vanderbilt Uni ; Divison of Nephrology, Nashville, Tennessee
  - Texas Transplant Inst., San Antonio, Texas
  - Uni of Texas Health Science Center At San Antonio; Organ Transplant Program, San Antonio, Texas
  - Uni of Washington Medical Center; Division of Allergy & Infectious Diseases, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital; Renal Transplant Unit, Camperdown, New South Wales
  - Monash Medical Centre; Renal Transplant Unit, Clayton, Victoria
  - Royal Melbourne Hospital; Nephrology, Parkville, Victoria
- Belgium (3):
  - Clin Univ de Bxl Hôpital Erasme, Brussels
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Brazil (5):
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
  - Hospital Israelita Albert Einstein; Intensive Care Unit, São Paulo, São Paulo
  - Faculdade de Medicina de Ribeirao Preto Usp; Campus Uni Rio, São Paulo, São Paulo
- Canada (4):
  - Uni of Alberta Hospital, Edmonton, Alberta
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Mcgill University - Royal Victoria Hospital; Oncology, Montreal, Quebec
- France (9):
  - Hopital Pellegrin; Departement Nephrologie, Bordeaux
  - Chu Grenoble - Hopital Albert Michallon; Departement de Cancero-Hematologie, Grenoble
  - Hopital Lapeyronie; Nephrologie, Montpellier
  - Hopital Hotel Dieu Et HME; Nephrologie Immunologie Clinique, Nantes
  - Ch Pitie Salpetriere; Urologie, Paris
  - Hopital Civil; Clinique Medicale, Strasbourg
  - CHU de Toulouse, Hopital Rangueil; Nephrologie-Tranplantation, Toulouse
  - Hopital Bretonneau; Nephrologie Transplantations, Tours
  - Hopitaux De Brabois; Nephrologie, Vandœuvre-lès-Nancy
- Germany (7):
  - Charité - Klinikum Mitte; Medizinische Klinik Für Nephrologie, Berlin
  - Charite - Campus, Virchow-Klinikum; Abteilung Fuer Nephrologie Und Intensivmedizin, Berlin
  - Universitätsklinikum Erlangen; Medizinische Klinik 4; Nephrologie und Hypertensiologie, Erlangen
  - Klinik Johann Wolfgang von Goethe Uni; Innere Medizin - Dialyse, Frankfurt
  - Med. Hochschule Hannover Zentrum Chirurgie Klinik f.Allgemein- Viszeral- und Transplantationschirur, Hanover
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Medizinische Klinik I, Lübeck
  - Klinikum der Universitaet Regensburg; Nephrologie, Regensburg
- Italy (4):
  - Policlinico di Bari; Divisione di Nefrologia, Dialisi e Trapianto, Bari, Apulia
  - POLICLINICO Universitatio A.Gemelli, Div. Chirurgia Generale e Trapianti d'Organo, Rome, Lazio
  - ASST GRANDE OSPEDALE METROPOLITANO NIGUARDA; Dipartimento di Nefrologia e Dialisi, Milan, Lombardy
  - Azienda Ospedaliera DI PADOVA; Divisione Malattie Infettive, Padua, Veneto
- Auckland City Hospital; Renal Unit, Level 15, Auckland, New Zealand
- Poland (3):
  - Collegium Medicum Uniwersytetu Jagielonskiego; Katedra I Klinika Nefrologii Cmuj, Krakow
  - Instytut Transplantologii A.M.; Klinika Medycyny Transplantacyjnej I Nefrologii, Warsaw
  - Akademia Medyczna Im. Piastow Slaskich; Klinika Nefrologii I Medycyny Transplantacyjnej, Wroclaw
- Romania (2):
  - Institutul de Urologie Si Transplant Renal Fundeni, Bucharest
  - Institutul de Urologie Si Transplant Renal Cluj Napoca, Cluj-Napoca
- Spain (6):
  - Hospital Universitari de Bellvitge; Servicio de Nefrologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Cruces; Servicio de Enfermedades Infecciosas, Barakaldo, Vizcaya
  - Hospital Universitari Vall d'Hebron; Servicio de Nefrologia, Barcelona
  - Hospital General Univ. Gregorio Maranon, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Enfermedades Infecciosas, Madrid
  - Hospital Universitario Dr. Peset; Servicio de Nefrologia, Valencia
- United Kingdom (10):
  - Antrim Hospital; Renal Dept, Antrim
  - Queen Elizabeth Hospital, Birmingham
  - SOUTHMEAD HOSPITAL; Richard Bright Dialysis Centre, Bristol
  - Western Infirmary; Division of Cardiovascular and Medical Sciences, Glasgow
  - Royal Liverpool Uni Hospital; Renal Dept, Liverpool
  - Royal London Hospital; Renal Unit, London
  - Manchester Royal Infirmary; Renal Transplant Unit, Manchester
  - Freeman Hospital; Nephrology, Newcastle upon Tyne
  - Nottingham City Hospital; Transplant Unit, Nottingham
  - Churchill Hospital; Oxford Transplant Center Renal Transplant Unit, Oxford

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Humar A, Lebranchu Y, Vincenti F, Blumberg EA, Punch JD, Limaye AP, Abramowicz D, Jardine AG, Voulgari AT, Ives J, Hauser IA, Peeters P. The efficacy and safety of 200 days valganciclovir cytomegalovirus prophylaxis in high-risk kidney transplant recipients. Am J Transplant. 2010 May;10(5):1228-37. doi: 10.1111/j.1600-6143.2010.03074.x. Epub 2010 Mar 26. PMID 20353469

RESULTS

PARTICIPANT FLOW:
Groups:
- Valganciclovir up to 100 Days: 900 mg valganciclovir orally daily for up to 100 days
- Valganciclovir up to 200 Days: 900 mg valganciclovir orally daily for up to 200 days
Period: Overall Study
Arm/Group | Valganciclovir up to 100 Days | Valganciclovir up to 200 Days
Started | 166 (Randomized) | 160 (Randomized)
Completed | 132 | 132
Not Completed | 34 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valganciclovir up to 100 Days | Valganciclovir up to 200 Days | Total
Number analyzed (Participants) | 164 | 156 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] — Safety population
  years | 48.5 (13.76) | 47.0 (13.51) | 47.8 (13.64)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety population
  Participants
    Female | 45 | 40 | 85
    Male | 119 | 116 | 235

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Developed Cytomegalovirus (CMV) Disease up to Month 12 Post-transplant
Description: Percentage of CMV-seronegative renal transplant recipients (R-) receiving a CMV-seropositive graft (D+) who developed CMV disease (confirmed and assumed) within 12 months post-transplant.
Time Frame: 12 months post-transplant
Population: Intent-to-treat population
Measure: Mean (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Valganciclovir up to 100 Days | Valganciclovir up to 200 Days
Number analyzed (Participants) | 163 | 155
Percentage of patients | 43.6 [35.8 to 51.5] | 23.9 [17.4 to 31.4]
Statistical Analysis 1: Comparison: Valganciclovir up to 100 Days vs Valganciclovir up to 200 Days; Test type: Superiority or Other; p <= 0.0002, Cochran-Mantel-Haenszel; Stratified by Center Pools; Odds Ratio (OR) = 0.40, 95% CI 2-sided [0.25 to 0.66]

2. Secondary Outcome: Percentage of Patients Who Developed CMV Disease up to Month 6 Post-transplant
Description: Percentage of CMV-seronegative renal transplant recipients (R-) receiving a CMV-seropositive graft (D+) who developed CMV disease (confirmed and assumed) within 6 months post-transplant.
Time Frame: 6 months post-transplant
Population: Intent-to-treat population
Measure: Mean (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Valganciclovir up to 100 Days | Valganciclovir up to 200 Days
Number analyzed (Participants) | 163 | 155
Percentage of patients | 36.2 [28.8 to 44.1] | 10.3 [6.0 to 16.2]
Statistical Analysis 1: Comparison: Valganciclovir up to 100 Days vs Valganciclovir up to 200 Days; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by Center Pools; Odds Ratio (OR) = 0.20, 95% CI [0.11 to 0.37]

3. Secondary Outcome: Percentage of Patients Who Developed CMV Disease up to Month 9 Post-transplant
Description: Percentage of CMV-seronegative renal transplant recipients (R-) receiving a CMV-seropositive graft (D+) who developed CMV disease (confirmed and assumed) within 9 months post-transplant.
Time Frame: 9 months post-transplant
Population: Intent-to-treat population
Measure: Mean (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Valganciclovir up to 100 Days | Valganciclovir up to 200 Days
Number analyzed (Participants) | 163 | 155
Percentage of patients | 43.6 [35.8 to 51.5] | 22.6 [16.3 to 30.0]
Statistical Analysis 1: Comparison: Valganciclovir up to 100 Days vs Valganciclovir up to 200 Days; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Stratified by Center Pools; Odds Ratio (OR) = 0.37, 95% CI [0.22 to 0.60]

4. Secondary Outcome: Percentage of Patients Who Developed CMV Disease up to Month 18 Post-transplant
Description: Percentage of CMV-seronegative renal transplant recipients (R-) receiving a CMV-seropositive graft (D+) who developed CMV disease (confirmed and assumed) within 18 months post-transplant.
Time Frame: 18 months post-transplant
Population: Intent-to-treat population
Measure: Mean (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Valganciclovir up to 100 Days | Valganciclovir up to 200 Days
Number analyzed (Participants) | 163 | 155
Percentage of patients | 47.9 [40.0 to 55.8] | 34.2 [26.8 to 42.2]
Statistical Analysis 1: Comparison: Valganciclovir up to 100 Days vs Valganciclovir up to 200 Days; Test type: Superiority or Other; p = 0.0126, Cochran-Mantel-Haenszel; Stratified by Center Pools; Odds Ratio (OR) = 0.56, 95% CI [0.35 to 0.88]

5. Secondary Outcome: Percentage of Patients Who Developed CMV Disease up to Month 24 Post-transplant
Description: Percentage of CMV-seronegative renal transplant recipients (R-) receiving a CMV-seropositive graft (D+) who developed CMV disease (confirmed and assumed) within 24 months post-transplant.
Time Frame: 24 months post-transplant
Population: Intent-to-treat population
Measure: Mean (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Valganciclovir up to 100 Days | Valganciclovir up to 200 Days
Number analyzed (Participants) | 163 | 155
Percentage of patients | 48.5 [40.6 to 56.4] | 34.2 [26.8 to 42.2]
Statistical Analysis 1: Comparison: Valganciclovir up to 100 Days vs Valganciclovir up to 200 Days; Test type: Superiority or Other; p = 0.0100, Cochran-Mantel-Haenszel; Stratified by Center Pools; Odds Ratio (OR) = 0.55, 95% CI [0.34 to 0.86]

ADVERSE EVENTS:
Description: Safety Population
Arm/Group | Valganciclovir up to 100 Days | Valganciclovir up to 200 Days
Serious Adverse Events (participants affected / at risk) | 94/164 | 78/156
Other Adverse Events (participants affected / at risk) | 133/164 | 141/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir up to 100 Days (N=164) | Valganciclovir up to 200 Days (N=156)
Cytomegalovirus Infection (Infections and infestations) | 21 | 5
Urinary Tract Infection (Infections and infestations) | 7 | 10
Cytomegalovirus Syndrome (Infections and infestations) | 12 | 1
Gastroenteritis (Infections and infestations) | 2 | 3
Pyelonephritis Acute (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 1 | 3
Pneumonia (Infections and infestations) | 1 | 2
Cytomegalovirus Viraemia (Infections and infestations) | 2 | 0
Wound Infection (Infections and infestations) | 1 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Bacterial Infection (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Campylobacter Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cytomegalovirus Colitis (Infections and infestations) | 1 | 0
Cytomegalovirus Hepatitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Escherichia Sepsis (Infections and infestations) | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Febrile Infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Klebsiella Infection (Infections and infestations) | 1 | 0
Lung Infection Pseudomonal (Infections and infestations) | 0 | 1
Mediastinitis (Infections and infestations) | 0 | 1
Perirectal Abscess (Infections and infestations) | 1 | 0
Pneumonia Streptococcal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Subcutaneous Abscess (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 4 | 2
Renal Impairment (Renal and urinary disorders) | 3 | 2
Haematuria (Renal and urinary disorders) | 1 | 1
Ureteric Obstruction (Renal and urinary disorders) | 1 | 1
Ureteric Stenosis (Renal and urinary disorders) | 1 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Renal Tubular Disorder (Renal and urinary disorders) | 0 | 1
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 1
Renal Vein Thrombosis (Renal and urinary disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Abdominal Pain (Gastrointestinal disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1
Impaired Gastric Emptying (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Transplant Rejection (Immune system disorders) | 11 | 8
Kidney Transplant Rejection (Immune system disorders) | 3 | 0
Food Allergy (Immune system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 9
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Bicytopenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 4
Chest Pain (General disorders) | 0 | 2
Impaired Healing (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Catheter Related Complication (General disorders) | 0 | 1
Catheter Site Discharge (General disorders) | 1 | 0
Multi-organ Failure (General disorders) | 1 | 0
Non-cardiac Chest Pain (General disorders) | 0 | 1
Oedema Peripheral (General disorders) | 0 | 1
Blood Creatinine Increased (Investigations) | 10 | 8
Lymphocele (Vascular disorders) | 2 | 3
Deep Vein Thrombosis (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 2 | 0
Phlebitis (Vascular disorders) | 2 | 0
Arterial Stenosis (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Iliac Artery Stenosis (Vascular disorders) | 1 | 0
Shock Haemorrhagic (Vascular disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 0 | 1
Complications of Transplanted Kidney (Injury, poisoning and procedural complications) | 2 | 1
Graft Dysfunction (Injury, poisoning and procedural complications) | 0 | 2
Complications of Transplant Surgery (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Medical Device Complication (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post Procedural Fistula (Injury, poisoning and procedural complications) | 1 | 0
Ureteric Anastomosis Complication (Injury, poisoning and procedural complications) | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Wound Secretion (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Acute Coronary Syndrome (Cardiac disorders) | 0 | 2
Arrhythmia (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 2
Angina Pectoris (Cardiac disorders) | 0 | 1
Arrhythmia Supraventricular (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Mitral Valve Disease (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0
Clonus (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Hereditary Haemorrhagic Telangiectasia (Congenital, familial and genetic disorders) | 0 | 1
Renal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Ureteral Stent Removal (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valganciclovir up to 100 Days (N=164) | Valganciclovir up to 200 Days (N=156)
Leukopenia (Blood and lymphatic system disorders) | 41 | 58
Anaemia (Blood and lymphatic system disorders) | 29 | 24
Neutropenia (Blood and lymphatic system disorders) | 22 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 8
Diarrhoea (Gastrointestinal disorders) | 41 | 48
Constipation (Gastrointestinal disorders) | 24 | 14
Nausea (Gastrointestinal disorders) | 18 | 17
Abdominal Pain (Gastrointestinal disorders) | 12 | 8
Vomiting (Gastrointestinal disorders) | 6 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 7 | 8
Dyspepsia (Gastrointestinal disorders) | 3 | 11
Urinary Tract Infection (Infections and infestations) | 20 | 29
Nasopharyngitis (Infections and infestations) | 17 | 12
Upper Respiratory Tract Infection (Infections and infestations) | 14 | 14
Oedema Peripheral (General disorders) | 35 | 30
Pyrexia (General disorders) | 17 | 10
Fatigue (General disorders) | 7 | 14
Hypophosphataemia (Metabolism and nutrition disorders) | 20 | 18
Hyperkalaemia (Metabolism and nutrition disorders) | 20 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 10
Tremor (Nervous system disorders) | 19 | 25
Headache (Nervous system disorders) | 16 | 9
Hypertension (Vascular disorders) | 21 | 19
Hypotension (Vascular disorders) | 10 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Insomnia (Psychiatric disorders) | 12 | 10
Blood Creatinine Increased (Investigations) | 11 | 9
Haematuria (Renal and urinary disorders) | 7 | 9
Rash (Skin and subcutaneous tissue disorders) | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.